CLINICAL TRIAL: NCT04785664
Title: Assessing the Impact of Community-based Pro-Active Monitoring Program (CAMP) on Community-dwelling Citizens Aged More Than 80
Brief Title: Community-based Pro-Active Monitoring Program (CAMP) and Older Adults
Acronym: CAMP-80
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Rome Tor Vergata (Other)
Collaborators: Comunità di S.Egidio ACAP Onlus (Unknown)
Responsible Party: Principal Investigator, Giuseppe Liotta, Associate Professor, University of Rome Tor Vergata
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: LLE001
Record Dates: First submitted 2021-02-01; First posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Social Isolation; Frailty
Keywords: Frail Elderly; Aged,80 and over; Social Isolation; Social Support; Mortality; Functional Geriatric Evaluation; Hospital Admission Rate
MeSH Terms: conditions — Social Isolation; Frailty

STUDY DESIGN:
Intervention Model Description: The study is a pragmatic trial according which, according to the ecological model, provides for a Community-based Pro-Active Monitoring intervention, on people aged>80, compared with a standard of care in two Italian Regions. The study is articulated in two phases: the baseline assessment provides a multidimensional assessment of the Functional Geriatric Evaluation questionnaire to the Long Live the Elderly (LLE) and Standard of Care (SoC) cohort. The follow up provides to collect information as Hospital Admission, Emergency Room accesses, Mortality rate, Admission to LCT facilities and use of home care services, with the collaboration of GPs and the regional database. The follow up will be gathered every six months over three years.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LLE- Long Live the Elderly! (Experimental): The group has been randomized among the "Long Live the Elderly!" (LLE) clients in two cities: Rome and Naples. The LLE central database includes all the participants to the program in Naples and Rome who have been administered the Functional Geriatric Evaluation (FGE) questionnaire.
  Interventions: Other: Community-based pro-Active Monitoring Program
- SoC- Standard of Care (No Intervention): No intervention will be carried out. The control group is selected by randomization from a pool of over-80s followed up by General Practitioners in the same cities who have been available to be involved in the study. Each GP provided a list of patients which 10 names have been selected from by randomization. The total pool consisted of approximately 8500 individuals. The sample was made up of 690 selected patients of which 83 (12.02%) refused to participate in the study.

INTERVENTIONS:
Other: Community-based pro-Active Monitoring Program — The Intervention provides phone monitoring addressed to all the clients and home visits tailored to the individual needs. Moreover, it activates other formal or informal care resources based on the needs of the patients reported in the Individualized Care Plan (ICP) which derives from the assessment of multidimensional frailty. The main peculiarity of the program is that the operators identify the main problem of the client and try to track down the best solution in agreement with the client. It can be a health or social intervention or a different kind. Interventions may include assistance to make clients' houses safer thereby reducing risk factors for falls or reviewing the therapeutic scheme to improve patient adherence to the treatment in collaboration with the GP.
  Arms: LLE- Long Live the Elderly!

SUMMARY:
Background: According to World Health Organization the world population is rapidly aging, and this impacts Health and Social Services. To improve older adults' quality of life and to reduce negative outcomes is necessary to provide appropriate care at affordable costs. To achieve this goal and to address the most effective intervention, stratification by frailty and negative outcomes is needed. Another crucial point to older adults is social isolation, this is related to the extension and quality of life of the individual's relationship network. Social isolation, as well as the level of frailty, are associated with an increased risk of death, hospitalization, and institutionalization.

Results: Analysis of data collected in the Lazio region during the pre-intervention phase is finished. Total patients enrolled are 1185 (578 cases and 607 control). The intervention is focused on increasing social capital at the individual and community level and aimed at improving survival among the cases as well as reducing the use of hospital and residential Long-Term Care.

Conclusions: The proposed study will address a crucial issue: assess the impact of a bottom-up care service consisting of social and health interventions aimed at reducing social isolation and improving access to health care services. The results of the study will be shared in the country, to reach the larger spread and to direct the policymaker.

Objective: The objective of this study is to evaluate the impact of a community-based proactive monitoring program. This study aims to improve community care by measuring the effect in countering the negative outcomes related to the frailty of older adults (over 80).

Methods: A prospective pragmatic trial will be carried out to describe the impact of an intervention on people aged>80, adjusted for relevant parameters: demographic variables, comorbidities, disability, and bio-psycho-social frailty. The multidimensional frailty will be evaluated with the Functional Geriatric Evaluation questionnaire that is a validated tool. The questionnaire was administrated at baseline to the two groups. Two clusters of patients have been enrolled and interviewed. The first made up of 578 cases (undergoing the intervention) and the second by 607 controls, among which no intervention will be performed. Case cluster intervention is a Community-based Pro-Active Monitoring Program performed by a multidisciplinary team on individual needs (level of frailty, social isolation, and physical disability). The primary outcome of this study is the evaluation of Mortality, Acute Hospital Admission rates, Emergency Room Visit rates, and Institutionalization rates. Data will be collected over three years in two cities: Rome and Naples.

ELIGIBILITY:
Inclusion Criteria:

* People enrolled into the study must be older than 80 years old
* People enrolled into the study had to answer to the FGE questionnaire.
* Advanced mental impairment was not an exclusion criteria, but in such cases the consent have been signed by the closest relative who also answered to the questionnaire on behalf of the selected participant.

Exclusion Criteria:

* People living in an institution (nursing homes or similar) have been excluded.

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1185 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of death | 3 years
  Mortality will be measured at 1 and 3 years from the collected data, it will be studied as a standardized rate adjusted for gender, age, and frailty level in LLE and SoC cohort. It will be the number of patient death per unit of time (1 year and 3 years).
Incidence of hospitalization | 3 years
  Hospitalization will be measured as a standardized rate (adjusted for gender, age, and frailty) in LLE and SOC groups at 1 year and 3 years (excluding patients transferred to another Region). Hospitalization will be measured on three factors: 1) the number of hospital admission for patients; 2) the number of hospitalization days; 3) the number of hospitalized patients.
Incidence of ER admission | 3 years
  Emergency Room admission will be measured in LLE and SoC cohort at 1 and 3 years (excluding patients transferred to another Region). ER, admission will be based on two indicators: 1) the number of ER admissions per patient; 2) the number of patients admitted to the ER.
Incidence of admission to LTC facilities | 3 years
  Admission to Long-Term- Care facilities will be measured as a standardized rate (adjusted for gender, age, and frailty) in LLE and SOC groups at 1 and 3 years. It will include the number of patients accessing LTC facilities per observation period.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rome Tor Vergata, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Liotta G, O'Caoimh R, Gilardi F, Proietti MG, Rocco G, Alvaro R, Scarcella P, Molloy DW, Orlando S, Mancinelli S, Palombi L, Stievano A, Marazzi MC. Assessment of frailty in community-dwelling older adults residents in the Lazio region (Italy): A model to plan regional community-based services. Arch Gerontol Geriatr. 2017 Jan-Feb;68:1-7. doi: 10.1016/j.archger.2016.08.004. Epub 2016 Aug 12. PMID 27567441
- [Result] Liotta G, Madaro O, Scarcella P, Inzerilli MC, Frattini B, Riccardi F, Accarino N, Mancinelli S, Terracciano E, Orlando S, Marazzi MC. Assessing the Impact of A Community-Based Pro-Active Monitoring Program Addressing the need for Care of Community-Dwelling Citizens aged more than 80: Protocol for a Prospective Pragmatic Trial and Results of the Baseline Assessment. Transl Med UniSa. 2020 Oct 31;23:22-27. doi: 10.37825/2239-9747.1004. eCollection 2020 Oct. PMID 33457318
- [Result] Liotta G, Scarcella P, Mancinelli S, Palombi L, Cancelli A, Marazzi MC. [The evaluation of care needs in elderly people: the use of Geriatric Functional Evaluation Questionnaire]. Ann Ig. 2006 May-Jun;18(3):225-35. Italian. PMID 16821500
- [Result] Liotta G, Inzerilli MC, Palombi L, Madaro O, Orlando S, Scarcella P, Betti D, Marazzi MC. Social Interventions to Prevent Heat-Related Mortality in the Older Adult in Rome, Italy: A Quasi-Experimental Study. Int J Environ Res Public Health. 2018 Apr 11;15(4):715. doi: 10.3390/ijerph15040715. PMID 29641436